CLINICAL TRIAL: NCT04427527
Title: Accelerating Colorectal Cancer Screening Through Implementation Science in Appalachia (ACCSIS)
Brief Title: Accelerating Colorectal Cancer Screening Through Implementation Science in Appalachia
Acronym: ACCSIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kentucky (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Ohio State University (Other)
Responsible Party: Principal Investigator, Mark Dignan, PhD, Professor, University of Kentucky
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Screening
Other Study IDs: 2018C0166; UH3CA233282 (NIH); 832127323 (Other: DUNS - The Ohio State University)
Record Dates: First submitted 2020-06-03; First posted 2020-06-11 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: Primary care clinics randomized to intervention or usual care
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Primary care clinics randomized to usual care do not receive intervention materials or attention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Multi-level Intervention (Experimental): Receives the project intervention first
  Interventions: Behavioral: Multi-level intervention to increase CRC screening
- Delayed Multi-level Intervention (No Intervention): Offered the intervention later in the project

INTERVENTIONS:
Behavioral: Multi-level intervention to increase CRC screening — Intervention for the community, providers, patients, clinics and systems
  Arms: Multi-level Intervention

SUMMARY:
This project aims to implement a multi-level group randomized trial, delayed intervention that includes components targeting clinics, providers, patients, and the community to increase colorectal cancer (CRC) screening, follow-up, and referral-to-care among patients age 50-74 in 12 counties in Appalachian Kentucky and Ohio. The 12 counties will be assigned to one of two study groups (early vs. delayed) and outcome measures (rate of CRC screening) will be obtained from clinic-level electronic health record data and a county-level behavioral assessment telephone survey. The hypothesis for the project is that the multi-level intervention will increase the clinic and county level CRC screening rates.

ELIGIBILITY:
Inclusion Criteria:

* age 50-74
* all races, sexes and genders
* resident of the study area

Exclusion Criteria:

.no exclusions based on gender, race or ethnicity

Ages: 50 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Self-report of gender
Enrollment: 5413 (Actual)
Dates: Start 2020-08-19 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
CRC screening - clinic level | 12 months
  Change in clinic-level screening rate from baseline to the end of the 12-month active intervention period, assessed through clinic electronic health record data

SECONDARY OUTCOMES:
CRC screening - community level | 12 months
  Self-reported participation in CRC screening from baseline to the end of the 12-month active intervention period, assessed through telephone surveys

CONTACTS AND LOCATIONS:
Overall Officials: Mark B Dignan, PhD, Principal Investigator — University of Kentucky
Locations (2):
- United States (2):
  - Markey Cancer Center, Lexington, Kentucky
  - Ohio State University, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: Yes
As outlined in the Notice of Award, each study site must make its Limited Data Set (LDS) accessible to other sites in the ACCSIS consortium. Information Management Services (IMS) will serve as the repository and have responsibility for creating a Limited Consolidated Data Set (LCDS) for analytic use of researchers both within and external to the ACCSIS consortium.
  Dataset Items in the LDS are defined by the Common Data Elements.
  There also will be a "public use data set" that consists of the Common Data Elements, available to external researchers. IMS will use a systematic process to remove identifiers.
  In addition, all data that underlie results in publications will be available per Notice of Award.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Baseline data available beginning 10/2020, follow-up data available 12/2023
Access Criteria: There are 2 classes of dataset requests: 1) public use and 2) special. Requestors submit necessary forms, including an agreement to acknowledge ACCSIS in publications and presentations. A public use data set containing common data elements will be made available to external researchers by application. IMS responds to public use dataset application by sending the requestor one-time access to a data download link. External researchers may also request a more customized data set. Requestors must first submit a brief concept form or ancillary studies form, for preliminary review by the ACCSIS Steering Committee (SC), before invitation to submit a full proposal. Full proposals receive review by NCI and Research Triangle Institute (RTI) before being forwarded to the SC for review and approval. Requestors report every 6 months on published articles or conference presentations to RTI. Requestors also are encouraged to make articles available through PubMed Central website.

REFERENCES:
- [Derived] Paskett ED, Kruse-Diehr AJ, Oliveri JM, Vanderpool RC, Gray DM, Pennell ML, Huang B, Young GS, Fickle D, Cromo M, Katz ML, Reiter PL, Rogers M, Gross DA, Fairchild V, Xu W, Carman A, Walunis JM, McAlearney AS, Huerta TR, Rahurkar S, Biederman E, Dignan M. Accelerating Colorectal Cancer Screening and Follow-up through Implementation Science (ACCSIS) in Appalachia: protocol for a group randomized, delayed intervention trial. Transl Behav Med. 2023 Sep 28;13(10):748-756. doi: 10.1093/tbm/ibad017. PMID 37202831
- [Derived] Kruse-Diehr AJ, Oliveri JM, Vanderpool RC, Katz ML, Reiter PL, Gray DM 2nd, Pennell ML, Young GS, Huang B, Fickle D, Cromo M, Rogers M, Gross D, Gibson A, Jellison J, Sarap MD, Bivens TA, McGuire TD, McAlearney AS, Huerta TR, Rahurkar S, Paskett ED, Dignan M. Development of a multilevel intervention to increase colorectal cancer screening in Appalachia. Implement Sci Commun. 2021 May 19;2(1):51. doi: 10.1186/s43058-021-00151-8. PMID 34011410

DOCUMENTS (1):
  • Informed Consent Form (2019-11-15): https://cdn.clinicaltrials.gov/large-docs/27/NCT04427527/ICF_000.pdf